CLINICAL TRIAL: NCT06310512
Title: Efficacy of Pharmacist Interventions Through the "Medication Therapy Management Pathway in Hypertensive Patients":A Prospective, Multicenter, Randomized, Controlled Study
Brief Title: Efficacy of Pharmacist Interventions Through the "Medication Therapy Management Pathway in Hypertensive Patients"
Acronym: PharmMTMH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Lin Yang, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ANZHEN HOSPITOL-LY-04
Record Dates: First submitted 2023-12-18; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Hypertension; Medication Therapy Management
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group patients will undergo structured drug treatment management at their first visit. During on-site follow-up at 1, 3, and 6 months, as well as telephone follow-up at the second week, 2 and 4 months, the patient's condition will be evaluated, corresponding information will be collected, and possible intervention measures will be taken for the patient.
  Interventions: Behavioral: Structured drug therapy management
- Non-Intervention group (No Intervention): For non intervention group patients, pharmacists evaluate the patient's condition and collect corresponding information at the first visit and on-site follow-up at 1, 3, and 6 months, explain the dosage and dosage of drugs to the patient, and remind them of medication contraindications. Necessary intervention measures are taken at the 6th month.

INTERVENTIONS:
Behavioral: Structured drug therapy management — Interventions mainly included (1) information collection, clinical assessment, and evaluation of medication regimens; (2) identification of and intervention for medication-related problems; (3) pharmacy instruction and education, and development of personal medication lists; and (4) follow-up and reassessment
  Arms: Intervention group

SUMMARY:
The goal of this Randomized Controlled Trial is to carry out in adult patients with primary hypertension whose blood pressure control is not up to standard. The main question it aims to answer are:

To explore the effect of pharmacists' implementation of "the medication therapy management pathway in hypertensive patients"on the patients with hypertension.

Participants will receive structured drug treatment management at the first diagnosis. During on-site follow-up in the first, third and sixth months, as well as telephone follow-up in the second week, second and fourth months, patients will be evaluated, corresponding information will be collected and possible interventions will be taken.

Researchers will compare the non intervention group to see if patients' blood pressure will also be reduced without intervention.

DETAILED DESCRIPTION:
The purpose of this study is to explore the effectiveness, safety, and cost-effectiveness of pharmacists implementing the Drug Treatment Management Pathway in the treatment of hypertension patients. This trial is a prospective, multi-center, randomized, controlled study. We plan to enroll 420 patients with primary hypertension who are over 18 years old and whose blood pressure control is not up to standard. Qualified participants who meet the inclusion and exclusion criteria were randomly divided into an intervention group of 280 cases and a non intervention group of 140 cases in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Outpatients diagnosed with primary hypertension who have not received treatment or are receiving antihypertensive medication;
3. Mild to moderate hypertensive patients with substandard blood pressure: home blood pressure >140/90 mmHg at least once in the last month or more, and the average sitting blood pressure in the clinic on the day of enrollment is >140/90 mmHg;
4. Expected survival > 12 months;
5. Voluntary participation in the trial and signing the informed consent form.

Exclusion Criteria:

1. Severe hypertension (mean SBP ≥180mmHg, or mean DBP ≥110mmHg), hypertensive emergency or hypertensive sub-emergency (systolic blood pressure >180 mmHg or diastolic blood pressure >120 mmHg);
2. Have a history or diagnosis of secondary hypertension, including but not limited to the following: renal hypertension, renal vascular hypertension, aortic stenosis, pheochromocytoma, Cushing's syndrome, cystic nephropathy, etc., but drug-induced hypertension is not an exclusion criterion;
3. Patients in the acute stage of the disease requiring emergency medical consultation;
4. patients with mental disorder, hearing impairment, intellectual disability, aphasia, etc., resulting in the inability to communicate or to comply with the study agreement
5. Patients with tumors;
6. Any other reasons that the investigator considers unsuitable for participation in the clinical trial that may affect the efficacy and safety evaluation of the study (including, but not limited to, the investigator's judgment that the subject lives far away and cannot be followed up as scheduled).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure | 6 months
  Change from baseline in mean seated systolic blood pressure at 6 months

SECONDARY OUTCOMES:
diastolic blood pressure | 6 months
  Changes from baseline in mean seated diastolic blood pressure at 6 months
Change from baseline in mean sitting systolic blood pressure at 3 months | 3 months
  Change from baseline in mean sitting systolic blood pressure at 3 months
Change from baseline in number of medication-related problems (MRP) at 6 months | 6 months
  Change from baseline in number of medication-related problems (MRP) at 6 months
Average number of medication-related problems (MRP) resolved after 6 months | 6 months
  Average number of medication-related problems (MRP) resolved after 6 months
The compliance rate of blood pressure after 6 months | 6 months
  The compliance rate of blood pressure after 6 months
Effective rate of blood pressure lowering after 6 months | 6 months
  Effective rate of blood pressure lowering after 6 months
Time to BP Attainment in Intervention and Non-Intervention Groups | From the date of enrollment to the date when the patient's first blood pressure meets the standard, the evaluation is conducted up to 6 months
  Time to BP Attainment in Intervention and Non-Intervention Groups
Changes from baseline in adherence scores at 6 months,the General Medication Compliance Scale (GMAS) was used. | 6 months
  The General Medication Compliance Scale (GMAS) was used, with a maximum score of 33 and a minimum score of 0. The higher the score, the higher the patient's compliance.
Economic indicators，mainly including the cost of implementing intervention measures and the impact of intervention measures on patient diagnosis and treatment costs | 6 months
  The implementation costs of intervention measures mainly include the development, installation, and annual maintenance costs of Interactive Network Response System (IWRS), labor costs of intervention measures, material costs incurred during the intervention process, multi center collaboration costs, and other costs incurred due to the intervention measures. Intervention measures have an impact on patient diagnosis and treatment costs, mainly including an increase in per visit outpatient expenses and medication costs.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lin, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No